CLINICAL TRIAL: NCT06486402
Title: An Observational Evaluation of Characteristics of Participants in Clinical
Brief Title: DISPARITY Study: An Observational Evaluation of Characteristics of Participants in Clinical Studies
Acronym: DISPARITY
Status: Active, not recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Prof. Dr. Marcus J. Schultz, Clinical Professor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: W23_111 # 23.136
Record Dates: First submitted 2024-03-26; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Participation Rate, Patient; Patient Participation
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: participation rate — participation rate

SUMMARY:
The aim of this study is to evaluate whether females are underrepresented in clinical studies in the Departments of Anaesthesia and Intensive Care, Amsterdam UMC, locations AMC and VUmc. The main outcome is Participation Prevalence Ratio (PPR), which means the representation of female/male patients in a study in relation to their representation in the disease population undergoing surgery.

To achieve this, we will use the average proportion of female participants enrolled per study and, in addition, data from the CBS for population benchmarking, determining the proportions of males and females undergoing surgery (elective cardiac and non-cardiac surgery) and the proportions of these populations in an academic hospital.

ELIGIBILITY:
Inclusion criteria:

* various clinical trials, both falling within and outside the scope of the Medical Research Involving Human Subjects Act
* adult patients undergoing various types of medical surgeries.

Exclusion criteria:

. studies which excluded or did not equally approach women beforehand

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study population consisted of various clinical trials, both falling within and outside the scope of the WMO, involving adult patients undergoing various types of medical surgeries. Importantly, only studies that did not preclude women beforehand and obtained consent before participation were included in the analysis.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Participation rate | 5 year
  Number of patients participating in a clinical trial

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided